CLINICAL TRIAL: NCT04005456
Title: LIFE-HOUSE: A Lifestyle Intervention and Functional Evaluation - a Health Outcomes Survey
Brief Title: Personalized Lifestyle Intervention for Improving Functional Health Outcomes Using N-of-1 Tent-Umbrella-Bucket Design
Acronym: LIFE-HOUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metagenics, Inc. (Industry)
Collaborators: Tufts Medical Center (Other); MetaProteomics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: LIFEHOUSE-PLMC
Record Dates: First submitted 2019-06-15; First posted 2019-07-02 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2022-04

CONDITIONS: Health, Subjective; Gastrointestinal Dysfunction; Cardiovascular Risk Factor; Autoimmune Diseases; Dental Diseases; Hormone Disturbance; Neurocognitive Dysfunction
Keywords: wellness; n-of-1 trial; detoxification; personalized medicine; functional medicine; 4P medicine; lifestyle medicine; homocysteine; dietary supplement; medical food; behavioral change; lifestyle modification; employee wellness program; functional capacity; food plan
MeSH Terms: conditions — Autoimmune Diseases; Stomatognathic Diseases; Endocrine System Diseases; Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (21):
- N of 1 Tent (Other): Personalized dietary supplements, food plans, and behavioral change support program for a broad group (both an employee population and those recruited from practitioner practices) inclusive of all study Participants and specifically generally healthy individuals, those with established disease/conditions requiring a personalized approach, those with diseases/conditions currently with low prevalence in our study population and those women currently pregnant or breastfeeding.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Wellness Umbrella (Other): Personalized dietary supplements, food plans, and behavioral change support program for a broad group of individuals characterized by minimal physical complaints and laboratory biomarkers of modest clinical significance.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Elevated Homocysteine Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for individuals from the Wellness Umbrella with elevated homocysteine level ≥ 10.4 µmol/L.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Dental Health Umbrella (Other): Personalized dietary supplements, food plans, and behavioral change support program for a broad group of individuals with established dental disease.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Immune Health Umbrella (Other): Personalized dietary supplements, food plans, and behavioral change support program for a broad group of individuals with autoimmune/inflammatory conditions (excluding metabolic disorders/atherosclerosis)
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Elevated Anti-Nuclear Antibodies (ANA) Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of individuals with elevated levels of antinuclear antibodies (preclinical symptomatology only).
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Autoimmune Conditions Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of individuals with an established diagnosis of an autoimmune conditions (Systemic Lupus Erythematosus, Rheumatoid Arthritis, Inflammatory Bowel Disease and Hashimoto's Thyroiditis) with ANA level >1:80 titer, rheumatoid factor (RF) ≥ 14 IU/ml, fecal calprotectin ≥ 50 mcg/g and thyroid autoantibody levels specifically thyroglobulin antibodies ≥ 115 IU/ml and/or thyroid peroxidase antibodies ≥ 35 IU/ml.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Symptomatic Fatigue/Myalgias Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for a broad employee health group with symptoms of persistent fatigue and myalgias.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Gastrointestinal Health Umbrella (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of individuals with conditions associated with issues of gastrointestinal health and of environmental toxicity or dysfunction related to detoxification of external toxins and internal metabolites.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Irritable Bowel Syndrome (IBS) Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of individuals with conditions associated with issues of gastrointestinal health.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Detoxification Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of individuals with conditions associated with issues of environmental toxicity or dysfunction related to detoxification of external toxins and internal metabolites.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Wellness Detoxification Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of individuals characterized by minimal physical complaints and normal biomarkers.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Metabolic Health Umbrella (Other): Personalized dietary supplements, food plans, and behavioral change support program for a broad group of participants classified as desirable weight with and without markers of dysglycemia/dyslipidemia or overweight/obese with and without markers of dysglycemia/dyslipidemia).
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Consequences of Metabolic (Dys)function Bucket C/S Design (Other): Personalized dietary supplements, food plans, and behavioral change support program for a broad group of participants classified as desirable weight with and without markers of dysglycemia/dyslipidemia or overweight/obese with and without markers of dysglycemia/dyslipidemia). C/S = crossover
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Consequences of Metabolic (Dys)function Bucket R/I Design (Other): Personalized dietary supplements, food plans, and behavioral change support program for a broad group of participants classified as desirable weight with markers of dysglycemia/dyslipidemia or overweight/obese with and without markers of dysglycemia/dyslipidemia). R/I = randomization/inclusion
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Ketogenic Product Development Exploratory Group (Other): Subgroup investigation in participants (classified as desirable weight with and without markers of dysglycemia/dyslipidemia or overweight/obese with and without markers of dysglycemia/dyslipidemia) during their 8- or 12-week ketogenic program intervention phase
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Reproductive Health Umbrella (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of participants with conditions associated with reproductive and hormonal health (including polycystic ovary syndrome, premenstrual syndrome, endometriosis, peri-menopause and menopausal conditions, women currently pregnant or breastfeeding, testosterone deficiency and andropause/late onset hypogonadism, and prostate health).
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Perimenopausal and Menopausal Transitions Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of women with conditions associated with reproductive and hormonal health specifically peri-menopause and menopausal conditions.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Premenstrual Syndrome Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of women with conditions associated with reproductive and hormonal health specifically premenstrual syndrome.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Polycystic Ovary Syndrome (PCOS) Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of women with PCOS with signs/symptoms/biomarkers of both metabolic dysfunction and hormonal derangements.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan
- Andropause/Late Onset Hypogonadism Bucket (Other): Personalized dietary supplements, food plans, and behavioral change support program for a group of men with conditions associated with reproductive and hormonal health specifically testosterone deficiency and andropause/late onset hypogonadism.
  Interventions: Dietary Supplement: Supplements and/or medical foods; Behavioral: Behavioral change support program; Other: Food plan

INTERVENTIONS:
Dietary Supplement: Supplements and/or medical foods — Personalized dietary supplementation (e.g., multivitamins/minerals, probiotics, specialized pro-resolving mediators, marine oil, vitamin D, hormone support, methylation support, protein drink, phytochemicals, neurocognitive support, targeted ingredients)
Behavioral: Behavioral change support program — Program to implement lifestyle and behavioral change according to individuals' need.
Other: Food plan — Personalized food plan (e.g., basic wellness food plan, cardiometabolic food plan, high protein high phytonutrient food plan, ketogenic food plan, detoxification food plan, anti-inflammatory food plan, neuro food plan)

SUMMARY:
The LIFE-HOUSE research project is designed to evaluate the impact of a personalized lifestyle intervention program on functional capacity as an approach to quantitating health, and its relationship to well understood disease risk determinants.

LIFE-HOUSE will utilize an innovative Tent-Umbrella-Bucket design.

Participants will gather under the Tent of an all-inclusive 'N of 1' Case Series providing a shelter of Functional Medicine interventions against the storm of chronic disease. Under this Tent are a collection of Umbrellas where participants with similar clinical challenges are evaluated as clinically defined groups with loose guidelines for the planned interventions. Finally, participants standing under these Umbrellas may step into specific Buckets that gather individuals with nearly identical clinical presentations into more formally described prescriptive randomized arms for intervention.

Individuals will be offered the opportunity to participate in all Umbrellas and Buckets for which they qualify. They may accept or reject participation in any Umbrella or Bucket and yet remain eligible for participation in the overall Tent.

DETAILED DESCRIPTION:
It has been suggested that the best medicine should value four principles (4P) - medicine should be personalized, predictive, preventative and participatory. This 4P Medicine will thus be personalized and patient centered with a focus on the person who has the disease and not the disease the person has. It will be predictive as it identifies the pre-clinical trend/decline towards illness sooner than onset of symptoms that herald the loss of function and health. It will be preventative as the information gathered should offer opportunities to modify these trajectories towards illness and finally it will be participatory as individuals will be intimately involved in the gathering of data to identify trends and in the application of lifestyle measures to improve their lives.

There is a significant unmet need to identify the value of a personalized lifestyle intervention program for improving functional health outcomes. Whereas disease is well understood from traditional pathology-based indices, health is less easily defined. Historically, healthy has been the default term that is applied to an individual who is not recognized as having a disease. This definition of health as the absence of disease has resulted in the delivery of health and wellness as often lying outside the purview of medicine.

An evolving definition of health, however, is to recognize that it is related to the functional capacity of the individual. Functional capacity can be categorized in four assessment areas: physiological, physical, cognitive and emotional. All four of these subcategories are quantifiable by both qualitative and quantitative metrics. The effects on health of a multi-modal personalized lifestyle medicine intervention program can best be evaluated by using functional determinants.

Functional Medicine is an integrative medicine philosophy that uniquely incorporates 4P Medicine with a focus on function and dysfunction and the necessity to consider the physiological events that determine the balance between the two. The LIFE-HOUSE research project is designed to evaluate the impact of a personalized lifestyle intervention program on functional capacity as an approach to quantitating health, and its relationship to well understood disease risk determinants.

Individuals will be offered the opportunity to participate in all Umbrellas and Buckets for which they qualify. They may accept or reject participation in any Umbrella or Bucket and yet remain eligible for participation in the overall Tent. Due to the structure of the uniquely defined yet overlapping system of Umbrellas and Buckets, a specific Subject may participate consecutively and/or sequentially in a series of Umbrella and Buckets as applicable and their data may be included in multiple Umbrella and Bucket analyses.

ELIGIBILITY:
General Inclusion Criteria for 'N of 1' Tent:

* male or female
* ages 18-80, inclusive
* willing to give written informed consent to participate in the study

General Exclusion Criteria for 'M of 1' Tent:

* Medical History and Concurrent Diseases:
* A serious, unstable illness including cardiac, hepatic, renal, gastrointestinal, respiratory, endocrinologic, neurologic, immunologic/rheumatological, or hematologic disease.
* Known infection with HIV, TB or Hepatitis B or C.
* Inability to comply with study and/or follow-up visits.
* Any concurrent condition (including clinically significant abnormalities in medical history, physical examination or laboratory evaluations) which, in the opinion of the PI, would preclude safe participation in this study or interfere with compliance.
* Any sound medical, psychiatric and/or social reason which, in the opinion of the PI, would preclude safe participation in this study or interfere with compliance.

The following describes specific inclusion and/or exclusion criteria applicable to individual study arms.

----------------------------------------------------------

Wellness Umbrella:

Specific Exclusion Criteria:

* MOS SF-36 QN general score < 60

Elevated Homocysteine Bucket:

Specific Inclusion Criteria:

* Elevated Homocysteine Level ≥ 10.4 µmol/L

Specific Exclusion Criteria:

* MOS SF-36 QN general score < 60

Dental Health Umbrella:

Specific Inclusion Criteria:

* Participants with extensive gingivitis/periodontitis/Caries/Painful teeth/Fractured Teeth. Identification of any of the following on physical exam: gingivitis, receding gumlines, periodontitis, fractured teeth, multiple unrestored caries. Identification on history of bleeding gums, bleeding while flossing, bleeding when brushing, chronic sores in the mouth, painful teeth, pain when biting on aluminum foil.

Neurological Health Umbrella:

Specific Inclusion Criteria:

* Elevated score on any subscale of Depression Anxiety Stress Scale (DASS) QN; and/or a score demonstrating mild or moderate depression or anxiety on Beck Depression Score and Beck Anxiety Score; and/or a MOS SF-36 subscale Emotional Role Functioning or Mental Health < 50; and/or PROMIS Cognitive Function QN score < 50.

Autoimmune and Inflammatory Conditions Umbrella:

Specific Inclusion Criteria:

* Symptoms, signs, laboratory biomarkers or diagnosis consistent with the features/diagnosis of an Autoimmune/Inflammatory Condition (excluding metabolic disorders/atherosclerosis) and ill-defined conditions characterized by symptomatic fatigue/myalgias.

Elevated ANA Bucket:

Specific Inclusion Criteria:

* General Inclusion Criteria for Autoimmune and Inflammatory Conditions Umbrella
* Elevated ANA Level > 1:40 titer (A specified sub-group for analysis will be all with two baseline elevated ANA Level > 1:40 titer.)

Specific Exclusion Criteria:

* Symptoms, signs, laboratory biomarkers (excluding ANA) or diagnosis consistent with the features/diagnosis of an Autoimmune/Inflammatory Condition (excluding metabolic disorders/atherosclerosis)

Autoimmune Conditions Bucket:

Specific Inclusion Criteria:

* Established Diagnosis of an autoimmune condition (Systemic Lupus Erythematosus, Rheumatoid Arthritis, Inflammatory Bowel Disease and Hashimoto's Thyroiditis) with ANA level >1:80 titer, rheumatoid factor (RF) ≥ 14 IU/ml, fecal calprotectin ≥ 50 mcg/g and thyroid autoantibody levels specifically thyroglobulin antibodies ≥ 115 IU/ml and/or thyroid peroxidase antibodies ≥ 35 IU/ml.

Symptomatic Fatigue and Myalgia Bucket:

Specific Inclusion Criteria:

* Two of the following five features have been generally present for at least 3 months:

  * Widespread bodily pain (pain in 3 of 5 regions (Left upper, right upper, left lower, right lower, axial) with and without symptomatic trigger points
  * Generalized fatigue
  * Sleep disturbances including awakening unrefreshed
  * Cognitive (memory or thought) problems
  * Post-exertional malaise

Gastrointestinal Health Umbrella:

Specific Inclusion Criteria:

* Symptoms, signs, laboratory biomarkers or diagnosis consistent with the features/diagnosis of Irritable Bowel Syndrome and other GI symptomatology (excluding Inflammatory Bowel Disease) as well as physiological challenges with healthy detoxification

IBS Bucket:

Specific Inclusion Criteria:

* Symptoms, signs, laboratory biomarkers or diagnosis consistent with the features/diagnosis of Irritable Bowel Syndrome and other GI symptomatology (excluding Inflammatory Bowel Disease)

Detoxification Bucket:

Specific Inclusion Criteria:

* Symptoms, signs, laboratory biomarkers or diagnosis consistent physiological challenges with healthy detoxification

Wellness Detoxification Bucket:

Specific Inclusion Criteria:

* Symptoms, signs, laboratory biomarkers or diagnosis consistent physiological challenges with healthy detoxification

Metabolic Health Umbrella:

Specific Inclusion Criteria:

* BMI>= 18.5 and <40

Consequences of Metabolic Function/Dysfunction Bucket - Crossover Design:

Specific Inclusion Criteria:

* BMI>= 18.5 and <40
* Metabolic Dysfunction is defined as having at least two of the following: Glucose ≥ 100 mg/dl; Homeostatic Model of Assessment for Insulin Resistance (HOMA-IR) (Glucose [mg/dl]Insulin [µiu/L)/405), score ≥ 2.0; HbA1c ≥ 5.7%; Triglycerides ≥ 100 mg/dl; Low Density Lipoprotein Particle Number (LDLp) >1000, lipoprotein (a) (lp(a)) > 30 mg/dl ; HDL (women) ≤ 50 ng/ml; HDL (men) ≤ 40 ng/ml; and blood pressure ≥ 135/85 mm Hg.

Specific Exclusion Criteria:

* Any of the following: Fasting Blood Glucose ≥ 125mg/dl; HbA1c ≥ 6.5% and Blood Pressure ≥ 165/95 mm Hg.

Consequences of Metabolic Function/Dysfunction Bucket - Randomization/Inclusion Design:

Specific Inclusion Criteria:

* BMI>= 18.5 and <40
* Metabolic Dysfunction is defined as having at least two of the following: Glucose ≥ 100 mg/dl; Homeostatic Model of Assessment for Insulin Resistance (HOMA-IR) (Glucose [mg/dl]Insulin [µiu/L)/405), score ≥ 2.0; HbA1c ≥ 5.7%; Triglycerides ≥ 100 mg/dl; Low Density Lipoprotein Particle Number (LDLp) >1000, lipoprotein (a) (lp(a)) > 30 mg/dl; HDL (women) ≤ 50 ng/ml; HDL (men) ≤ 40 ng/ml; and blood pressure ≥ 135/85 mm Hg

Specific Exclusion Criteria:

* Any of the following: Fasting Blood Glucose ≥ 125mg/dl; HbA1c ≥ 6.5% and Blood Pressure ≥ 165/95 mm Hg.

Reproductive Health Umbrella:

Specific Inclusion Criteria:

* Applicable to female Participants: a clinical diagnosis of fibrocystic breast and/or increased risk for Breast cancer, polycystic ovary syndrome, endometriosis, premenstrual syndrome, peri-menopause and menopausal conditions.
* Applicable to male Participants: a diagnosis of testosterone deficiency and andropause/late onset hypogonadism or prostate health concerns.

Perimenopausal and Menopausal Transitions Bucket:

Specific Inclusion Criteria:

* Female with signs/symptoms consistent with a clinical diagnosis of peri-menopause and menopausal conditions.

Premenstrual Syndrome Bucket:

Specific Inclusion Criteria:

* Female with a diagnosis of premenstrual syndrome and/or signs/symptoms/biomarkers consistent with estrogen/progesterone imbalances.

PCOS Bucket:

Specific Inclusion Criteria:

* Female with signs/symptoms/biomarkers consistent with a clinical diagnosis of PCOS.

Andropause/Late Onset Hypogonadism Bucket:

Specific Inclusion Criteria:

* Male with signs/symptoms/biomarkers consistent with a clinical diagnosis of Andropause/Late Onset Hypogonadism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Employee health program inclusive of all gender and non-binary descriptions.
Enrollment: 400 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study Short Form 36 (MOS SF-36) questionnaire | Change from baseline at 12 months
  The MOS SF-36 is an indicator of overall health status. It has an eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability.
University of Rhode Island Change Assessment (URICA) questionnaire | Change from baseline at 12 months
  URICA questionnaire is a 32 item self-report measure that includes 4 subscales measuring the stages of change: Precontemplation, Contemplation, Action, and Maintenance (there is also a 24 item version). Responses are given on a 5 point Likert scale ranging from (1=strong disagreement to 5=strong agreement),
Depression Anxiety, Stress Scale (DASS) questionnaire | Change from baseline at 12 months
  The Depression, Anxiety and Stress Scale is a 21 items questionnaire that includes a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Outcome is divided into normal, mild, moderate, severe, and very severe for each of the 3 categories: Depression, Anxiety, and Stress. A low score represents the normal and the higher the score the more severe the outcome.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Change from baseline at 12 months
  BMI is measured in (weight in kilogram (kg)/ height in meter (m)^2) outcome in double digits.
Waist Circumference (WC) | Change from baseline at 12 months
  WC is measured in centimeters (cm)
Hip Circumference (HC) | Change from baseline at12 months
  HC is measured in cm
Waist to Hip Ratio (WHR) | Change from baseline at 12 months
  WHR is numerical (0.00) and is and indicator for major health risk.
Height | Change from baseline at 12 months
  Height in meter (m)
Weight | Change from baseline at12 months
  Weight in kilogram (kg)
Glucose | Change from baseline at 12 months
  Fasting glucose levels measured in blood in milligram/deciLiter (mg/dL)
Total Cholesterol | Change from baseline at 12 months
  Fasting total cholesterol level is measured in serum in mg/dL
Anti-Nuclear Antibodies (ANA) | Change from baseline at 12 months
  ANA is measured as a titer by serum dilution detects autoimmune disease.
25-hydroxy (OH) Vitamin D3 | Change from baseline at 12 months
  25-OH Vitamin D3 is measured in blood in nanogram/milliLiter (ng/mL) detects deficiencies.
High sensitivity C-Reactive Protein (Hs-CRP) | Change from baseline at 12 months
  Hs-CRP is measured in blood in mg/L detects inflammation.
Homocysteine | Change from baseline at 12 months
  Homocysteine is measured in serum in micromol/Liter (µmol/L)
Omega-3 Fatty Acids | Change from baseline at 12 months
  Omega-3 fatty acids: Eicosapentaenoic (EPA), Docosahexaenoic (DHA), and Docosapentaenoic (DPA) levels are measured in % weight.
Beck Depression Inventory (BDI) | Change from baseline at 12 months
  BDI is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. Rating system: 1-10: These ups and downs are considered normal; 11-16: Mild mood disturbance; 17-20: Borderline clinical depression; 21-30: Severe depression; over 40: Extreme depression
Beck Anxiety Inventory (BAI) | Change from baseline at12 months
  BAI is a multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults.The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs[4] are:
  0-7: minimal anxiety 8-15: mild anxiety 16-25: moderate anxiety 26-63: severe anxiety
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Test | Change from baseline at 12 months
  PROMIS Sleep Disturbance Test is a self-scored test to identify sleep disturbance. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance. The T-scores are interpreted as follows: Less than 55 = None to slight 55.0-59.9 = Mild 60.0-69.9 = Moderate 70 and over = Severe
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Test | Change from baseline at12 months
  PROMIS Anxiety test is a 7-item questionnaire that assesses the pure domain of anxiety in individuals age 18 and older. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety. The T-scores are interpreted as follows: Less than 55 = None to slight 55.0-59.9 = Mild 60.0-69.9 = Moderate 70 and over = Severe
Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form (SF) | Change from baseline at 12 months
  PROMIS Depression SF is an 8-item questionnaire that assesses the pure domain of depression in individuals age 18 and older. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.The T-scores are interpreted as follows: Less than 55 = None to slight 55.0-59.9 = Mild 60.0-69.9 = Moderate 70 and over = Severe

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lamb, MD, Principal Investigator — Personalized Lifestyle Medicine Center
Locations (1):
- Personalized Lifestyle Medicine Center, Gig Harbor, Washington, United States

IPD SHARING:
Plan to Share IPD: No